CLINICAL TRIAL: NCT03813706
Title: Prospective Study for the Dissection of Lymph Node Posterior to Right Recurrent Laryngeal Nerve for Papillary Thyroid Carcinoma
Brief Title: the Dissection of Lymph Node Posterior to Right Recurrent Laryngeal Nerve for Papillary Thyroid Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Luo Dingcun, vice president of hospital, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangU20190115
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Lymph Node Metastases
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LN-prRLN dissection (Active Comparator)
  Interventions: Procedure: lymph node dissection
- no LN-prRLN dissection (Experimental)
  Interventions: Procedure: lymph node dissection

INTERVENTIONS:
Procedure: lymph node dissection — The right cervical central compartment VI is subdivided into right cervical central VI-1 subzone and VI-2 subzone. Right central VI-1 subzone lies anterior to the RLN bounded by the hyoid bone superiorly, the suprasternal notch inferiorly, the inner edge of the common carotid artery laterally, and the midline of the trachea medially. Right central VI-2 subzone lies posterior to the right RLN. The superior, inferior, lateral, and medial borders are the laryngeal entry points of RLN, the intersection of the RLN with the innominate artery (near the right apical pleura), the inner edge of the common carotid artery, and esophagus, respectively. The floor of right central VI-2 is the prevertebral fascia.

SUMMARY:
This study was completed in two stages. In the first stage, 2000 participants were enrolled according to the criteria. Following the principle of informed consent and voluntary consent of patients, the standard operation was "right or bilateral thyroidectomy + isthmus resection + right area VI lymph node dissection + left area VI lymph node dissection + lateral neck lymph node dissection". The age of participants, the size of right thyroid tumors, the invasion of the capsule and the number of lateral neck lymph node metastasis were counted to validate and improve the predictive model of lymph node posterior to the right recurrent laryngeal nerve in papillary thyroid cancer (Y=-0.029×age+0.771×tumor size+0.660×capsular invasion+1.331×right lateral lymph node metastasis-1.687, Y ≥0.16 means right recurrent laryngeal nerve posterior lymph node metastasis).

In the second stage, 2000 participants assessed by the model without posterior right recurrent laryngeal nerve metastasis were randomly divided into experimental group and control group according to the principle of informed consent and voluntary. The right recurrent laryngeal nerve posterior lymph nodes were not dissected in experimental group, while the right recurrent laryngeal nerve posterior lymph nodes were routinely dissected in control group. Through long-term follow-up and comparison of RFS and OS between the two groups, the investigators can scientifically evaluate the effectiveness of the "prediction model of lymph node posterior to right recurrent laryngeal nerve metastasis in papillary thyroid carcinoma", and seek evidence for accurate treatment of lymph node posterior to the right recurrent laryngeal nerve in thyroid papillary carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Phase I:

  1. aged from 18 years old to 80 years old;
  2. the primary treatment of patients with right or bilateral PTC;
  3. patients will voluntarily enter the study after informed consent.

Phase II:

1. aged from 18 years old to 80 years old;
2. the primary treatment of patients with right or bilateral PTC predicted to have no LN-prRLN metastasis by the "prediction model of LN-prRLN";
3. patients will voluntarily enter the study after informed consent.

Exclusion Criteria:

1. patients refused to participate in the study;
2. non first operation patients;
3. other malignant tumor history;
4. distant metastasis;
5. history of neck trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of thyroid cancer | Participants will be followed from the operation to 20 year (maximum)